CLINICAL TRIAL: NCT06039566
Title: A Trial Evaluating the Impact of N-acetylcysteine on Opioid Use in Patients Undergoing a Hysterectomy Procedure
Brief Title: NAC vs Placebo on Opioid Use for Hysterectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sylvia Wilson, Professor of Anesthesiology, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00130489
Record Dates: First submitted 2023-08-25; First posted 2023-09-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hysterectomy
Keywords: hysterectomy
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Placebo (Placebo Comparator): Patients will receive: Placebo 0 mg/kg (placebo: 0.45% NaCl or D5W) through an IV that will run for 60 minutes at the start of the procedure.
  Interventions: Drug: IV Placebo
- IV N-acetylcysteine (Active Comparator): Patients will receive: N-acetylcysteine (NAC) 150 mg/kg (Max dose 15,000 mg) through an IV that will run for 60 minutes at the start of the procedure.
  Interventions: Drug: IV N-acetylcysteine

INTERVENTIONS:
Drug: IV N-acetylcysteine — N-acetylcysteine (NAC) 150 mg/kg (Max dose 15,000 mg) through an IV that will run for 60 minutes at the start of the procedure
  Other Names: NAC
  Arms: IV N-acetylcysteine
Drug: IV Placebo — Placebo 0 mg/kg (placebo: 0.45% NaCl or D5W) through an IV that will run for 60 minutes at the start of the procedure.
  Other Names: Placebo
  Arms: IV Placebo

SUMMARY:
This study will enroll females who are ages 18 and older undergoing a laparoscopic or robotic, partial or full hysterectomy. Participants will be randomized to receive IV n-acetylcysteine or placebo during the first 60 minutes of their procedure. At various time points after the procedure patients will be asked to report their pain scores, and any pain medication taken.

ELIGIBILITY:
Inclusion

* Undergoing elective laparoscopic or robotic, full, or partial hysterectomy procedure
* 18 years of age and older

Exclusion

* Less than 40kg in weight
* Unable to provide written, informed consent
* History of an adverse or anaphylactoid reaction to acetylcysteine
* Active asthma, wheezing, or using inhaled bronchodilators
* Non-English speaking
* Insulin dependent diabetes if D5W is required
* Blood clotting disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 240 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption 0-72 hours post-study medication | 0-72 hours after study medication
  72-hour post-medication opioid consumption.

SECONDARY OUTCOMES:
Pain Scores | Study medication start to 72 hours post-study medication
  Using a Visual Analog Scale from 0-100, patients will report pain scores from 0-72 hours post-medication. A lower pain score means a better outcome.

OTHER OUTCOMES:
intraoperative opioid consumption | during the procedure (up to 12 hours)
  Total morphine milligram equivalents administered during the procedure
postoperative anesthesia care unit (PACU) opioid consumption | PACU Arrival until PACU Discharge up to 52 weeks
  Total morphine milligram equivalents administered in the PACU
non-opioid analgesic administration | Anesthesia start until PACU discharge up to 52 weeks
  Total other pain medication administered during the procedure and in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Wilson, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No